CLINICAL TRIAL: NCT05463081
Title: Clinical Trial of the Safety and Efficacy of Medical Device "Laser Medical Device "Magic Gyno""
Brief Title: Clinical Trial of "Magic Gyno" Laser Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MeLSyTech, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTMGLD-2022
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Female Urogenital Diseases; Urinary Incontinence; Prolapse Genital; Menopausal Syndrome; Postmenopausal Period; Vaginal Atrophy; Vaginal Prolapse; Postpartum Period; Sexual Dysfunction; Preoperative Care; Postoperative Care
Keywords: Laser; Vaginal; Neodymium Laser; Laser Treatment; Nanosecond; Female Urogenital Diseases; Pelvic Organ Prolapse
MeSH Terms: conditions — Female Urogenital Diseases; Urinary Incontinence; Uterine Prolapse; Sexual Dysfunction, Physiological; Pelvic Organ Prolapse | interventions — Laser Therapy; Hematologic Tests; Vaginal Smears

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genitourinary disorder (Experimental): Participants with:
  * stress urinary incontinence,
  * mixed urinary incontinence with a predominance of the stress component,
  * genitourinary menopausal syndrome,
  * dystrophic and atrophic processes in the genital area,
  * scleroatrophic changes in the urogenital region.
  Laser treatment of the vagina, vulva, and paraurethral region with "Magic Gyno" laser. In total, three procedures will be performed with an interval of 4 weeks.
  During the procedure, the following sequence of actions will be performed:
  1. st Stage - vaginal processing with a conical mirror handpiece,
  2. nd Stage - vaginal processing with a corner mirror handpiece,
  3. d Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.
  Interventions: Device: Laser treatment; Diagnostic Test: Blood test; Diagnostic Test: Clinical urine test; Diagnostic Test: Vaginal smear; Diagnostic Test: Pelvic ultrasound; Other: Female Sexual Function Index; Other: International Consultation on Incontinence Questionnaire - Short Form; Other: The Short Form Health Survey; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Vital signs determination; Diagnostic Test: pH of vagina determination; Diagnostic Test: Physical parameters determination
- Relaxation of vagina (Experimental): Participants with:
  * prolapse of the genitals I-II degree,
  * vaginal relaxation syndrome,
  * postpartum recovery,
  * sexual dysfunctions,
  * restoration of tone, turgor and tissue density of the urogenital area (Intimate rejuvenation, correction of age-related changes),
  * preoperative preparation for genital prolapse surgery and postoperative rehabilitation.
  Laser treatment of the vagina, vulva, and paraurethral region with "Magic Gyno" laser. In total, three procedures will be performed with an interval of 4 weeks.
  During the procedure, the following sequence of actions will be performed:
  1. st Stage - vaginal processing with a conical mirror handpiece,
  2. nd Stage - vaginal processing with a corner mirror handpiece,
  3. d Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.
  Interventions: Device: Laser treatment; Diagnostic Test: Blood test; Diagnostic Test: Clinical urine test; Diagnostic Test: Vaginal smear; Diagnostic Test: Pelvic ultrasound; Other: Female Sexual Function Index; Other: International Consultation on Incontinence Questionnaire - Short Form; Other: The Short Form Health Survey; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Vital signs determination; Diagnostic Test: pH of vagina determination; Diagnostic Test: Physical parameters determination

INTERVENTIONS:
Device: Laser treatment — Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 ns, the pause between pulses is 30 us. The energy of one pulse is about 1 mJ.
  General laser radiation parameters for 1st and 2nd stages are: beam with diameter of 4 millimeters (mm) scans treatment area by 4 circles with step of 2 mm (50 percentage (%) overlap), average power of 10-25 Watt (W), treatment time in one point of 1-10 seconds (s), treatment step of 5 mm, from 1 to 5 repetitions of total vagina treatment. General laser radiation parameters for 3d stage are: beam diameter of 6 mm, average power of 15-30 W, duration of ns-pulses packet of 50-100 milliseconds (ms), pause between packets of 50-100 ms, treatment duration up to 65 s, treatment in permanent motion with speed of 10-50 mm/s.
  The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.
Diagnostic Test: Blood test — Taking blood from a vein for Wassermann reaction (WR), human immunodeficiency viruses (HIV), hepatitis B infection (HBsAg), hepatitis C infection (HCVAg) determination, glucose test (to include the participant in the study) and clinical blood analysis (to include the participant in the study and evaluate procedure efficiency)
Diagnostic Test: Clinical urine test — Urine sampling for Clinical urine test (to include the participant in the study).
Diagnostic Test: Vaginal smear — Vaginal smear for flora investigation (to include the participant in the study and evaluate procedure efficiency)
Diagnostic Test: Pelvic ultrasound — Pelvic ultrasound investigation to determine pathologies of the pelvic through a gynecological probe (to include the participant in the study).
Other: Female Sexual Function Index — Female Sexual Function Index will be used to collect feedback on changes in the participants life quality (to evaluate procedure efficiency).
Other: International Consultation on Incontinence Questionnaire - Short Form — International Consultation on Incontinence Questionnaire will be used to collect feedback on changes in the participants' life quality (to evaluate procedure efficiency).
Other: The Short Form Health Survey — The Short Form Health Survey will be used to collect feedback on changes in the participants' life quality (to evaluate procedure efficiency).
Diagnostic Test: Vaginal Health Index — Vaginal Health Index will be investigated by clinical examination for vaginal elasticity, vaginal secretions, epithelial mucous membrane, vaginal hydration. Potential of hydrogen (pH) will be investigated by test-lines paper (to evaluate procedure efficiency).
Diagnostic Test: Vital signs determination — Vital signs determination (respiration rate, blood pressure, pulse rate, body temperature).
Diagnostic Test: pH of vagina determination — Potential of hydrogen (pH) of vagina will be investigated by test-lines paper (to evaluate procedure efficiency).
Diagnostic Test: Physical parameters determination — Physical parameters determination (body weight, age, height, body mass index).

SUMMARY:
The aim of this prospective study is investigation of efficiency and safety of medical device "Magic Gyno" in accordance with the stated purpose. To assess the condition of the vaginal walls and vulva before and after laser treatment, the following methods will be used: gynecology examination, vaginal health index, clinical blood test, vaginal flora examination, vaginal pH. International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF), Female Sexual Function Index (FSFI) and The Short Form Health Survey (SF-36) will be used to collect feedback on changes in the participants life quality. Total up to 70 participants with pathology of pelvic organs will be involved in the study. Participants will be divided into two groups: group with genitourinary symptoms and group with vaginal relaxation symptoms, by 35 participants in each. The time intervals between tests will be the same for both groups. The main hypothesis of the study is improvement in condition of the vaginal walls after laser treatment compared with the condition before treatment.

DETAILED DESCRIPTION:
The principle of participant distribution into groups is the character of vaginal walls and vulva pathology. Total up to 70 participants will be involved in the study. Participants will be divided into two groups: group with genitourinary symptoms and group with vaginal relaxation symptoms by 35 participants in each.

The types of examination of each group are the same and include:

General methods: demographic data determination, vital signs determination, gynecological examination, physical examination, clinical blood analysis with glucose determination, clinical urine test, vaginal smear for flora and oncocytology, pelvic ultrasound.

Special methods: vaginal smear for flora, vaginal pH determination, filling out the questionnaire (Female Sexual Function Index, International Consultation on Incontinence Questionnaire - Short Form, The Short Form Health Survey), Vaginal Health Index determination.

The treatment procedure of this study is the laser treatment of the vagina and vulva with a "Magic Gyno" laser with subsequent monitoring.

Treatment Technique:

Laser treatment procedure will be carried out in three stages. In total, three procedures will be performed with an interval of 4-6 weeks. One follow-up visit will follow: 90 days after the last procedure.

During the procedure, the following sequence of actions will be performed:

1. st Stage - vaginal processing with a conical mirror handpiece,
2. nd Stage - vaginal processing with a corner mirror handpiece,
3. rd Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.

Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 nanoseconds (ns), the pause between pulses is 30 microseconds (us). The energy of one pulse is about 1 millijoule (mJ). The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.

Participants of all groups will be tested with the general methods necessary to include the participant in the study at the first visit.

For both group: Studies will be carried out using special methods and then laser treatment of the vagina and vulva and paraurethral region will be performed during the 2nd, 3d, and 4th visits. Studies with all special methods will be performed during the 1st (to include participant in the study), 2nd (before the first treatment), 4th (before the last treatment) and 5th (90 days after the last treatment) visits.

Thus, direct comparison between participants condition before and 90 days after treatment within each group will be carried out.

The study will be carried out with the participation of Tver State Medical Academy.

All data obtained during the study will be transferred to the manufacturer of "MeLSyTech" Ltd.

The study will be monitored by "MeLSyTech" Ltd as follows:

In the start of study to ensure awareness of researchers about the plan, the rules for filling in case research forms, work with the device.

Once a 3 month, monitoring of provided documents (copies of individual registration records of participants (case research forms), informed consent, test results) for the complete filling of the forms; the clarity of filling out forms, the possibility of systematizing information from the forms of their assessment. Monitoring will be conducted with a coordinator visit of the research center and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

In the end of study monitoring will be conducted with a coordinator visit of the research center and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. The investigator submits a clinical evaluation report to the sponsor.

Statistics The analysis will be carried out within groups at different time intervals (analysis of matched groups).

Before performing statistical analysis of the data, the distribution type of the variables will be assessed. To assess the normality of distribution for each variable, histograms of frequency distributions will be visually evaluated, indicators of skewness, kurtosis, and the D'Agostino-Pearson normality test will be used.

In addition to checking the type of distribution of variables, the equality of variances of the studied groups will be assessed using the methods of analysis of variance, in particular the Brown-Forsythe test.

Methods of descriptive analysis will be used depending on the type of distribution of the variable. With a normal distribution, the mean (M) and standard deviation (SD) will be calculated. In case of an nongaussian distribution, the median (Me) and interquartile range will be calculated. Different algorithms of statistical analysis will be applied depending on the type of distribution of variables.

Comparison of the paired groups with a normal distribution, in case of the equality of the variances, will be carried out by the methods of analysis of variance ANOVA. Comparison of groups in pairs will be performed using the post-hoc method of posterior multiple comparisons (Tukey test).

Comparison of groups in which variables do not follow the normal distribution will be carried out using the methods of nonparametric analysis of variations: the Friedman test for matched groups.

Differences will be considered statistically significant if the significance P values are <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 years old in conditions caused by collagen deficiency in the treated area, women in premenopause and menopause;
* Participants who signed informed consent and fully informed about the purpose of the study;

Following disorders:

* Stress urinary incontinence,
* Mixed urinary incontinence with a predominance of the stress component,
* Genitourinary menopausal syndrome,
* Dystrophic and atrophic processes in the genital area,
* Scleroatrophic changes in the urogenital region,
* Prolapse of the genitals I-II degree,
* Vaginal relaxation syndrome,
* Postpartum recovery,
* Sexual dysfunctions,
* Restoration of tone, turgor and tissue density of the urogenital area (Intimate rejuvenation, correction of age-related changes),
* Preoperative preparation for genital prolapse surgery and postoperative rehabilitation.

Exclusion Criteria:

* Age up to 18 years;
* Inability or unwillingness to give informed consent to participate in a trial or to fulfill the requirements of a clinical trial;
* The presence of contraindications to the use of a medical device;
* Pregnancy;
* Bleeding disorders accompanied by a violation of blood clotting;
* Use of anticoagulant medicines (post-infarction and post-stroke conditions);
* Autoimmune diseases;
* Emerging infection diseases of any etiology;
* Damage to the skin (mucous membranes) in the area of laser treatment;
* Oncological diseases, cancer alertness;
* Decompensated diabetes;
* Photosensitizing drug administration;
* Decompensated somatic diseases;
* Decompensated cardiovascular disease, and other decompensated common diseases;
* Severe somatic diseases (heart failure, chronic renal failure, hepatitis, liver cirrhosis);
* Severe autoimmune diseases (including hemorrhagic vasculitis);
* Immunodeficiency (including HIV infection and AIDS);
* Severe mental and neurological disorders;
* Bedridden and immobile patients;
* COVID 19;
* Acute inflammatory diseases of the urogenital area;
* Acute purulent processes of the urogenital region;
* Bleeding of a natural nature (menstruation) and any other types of bleeding in the urogenital area;
* Postoperative scars up to 6 months;
* Lateral cysts of the vagina;
* Growing uterine fibroid;
* Fillers / suture in the area of laser exposure;
* The presence of varicose veins of the urogenital region and dilated capillary plexuses of the mucosa.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline of Vaginal Health Index Score | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Vaginal Health Index will be investigated by clinical examination for vagina:
  A. Vaginal elasticity (Characteristic=Points: None=1, Poor=2, Fair=3, Good=4, Excellent=5), B. Vaginal secretions (None=1; Sсant, thin yellow=2; Superficial, thin white=3; Moderate, thin white=4; Normal (white)=5), C. Epithelial mucous membrane (Petechiae noted before contact=1, Bleeding with light contact=2, Bleeds with scraping=3, Not friable thin epithelium=4, Normal=5), D. Vaginal hydration (None, surface inflamed=1, None, surface nod inflamed=2, Minimal=3, Moderate=4, Normal=5), E. pH will be investigated by test-lines paper (≥6.1=1, 5.6-6.0=2, 5.1-5.5=3, 4.7-5.0=4, ≤4.6=5).
  Score=A+B+C+D+E

SECONDARY OUTCOMES:
Mean Change from Baseline of "Desire" Score on the Female Sexual Function Index Questionnaire | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants answer questions:
  Q1. Over the past 4 weeks, how often did you feel sexual desire or interest? Answers = Points: almost always or always (5), most times (more than half the time) (4), sometimes (about half the time) (3), a few times (less than half the time) (2), almost never or never (1).
  Q2. Over the past 4 weeks, how would you rate your level (degree) of sexual desire or interest? Answers = Points: very high (5), high (4), moderate (3), low (2), very low or none at all (1)
  Score = (Score to Q1 + Score to Q2)x0.6
Mean Change from Baseline of "Arousal" Score on the Female Sexual Function Index Questionnaire | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants answer questions: Q3. Over the past 4 weeks, how often did you feel sexually aroused during sexual activity or intercourse? Q6. Over the past 4 weeks, how often have you been satisfied with your arousal (excitement) during sexual activity or intercourse? Answers = Points (Q3 and Q6): no sexual activity (0), almost always or always (5), most times (4), sometimes (3), a few times (2), almost never or never (1) Q4. Over the past 4 weeks, how would you rate your level of sexual arousal during sexual activity or intercourse? Answers = Points: no sexual activity (0), very high (5), high (4), moderate (3), low (2), very low or none at all (1) Q5. Over the past 4 weeks, how confident were you about becoming sexually aroused during sexual activity or intercourse? Answers=Points: no sexual activity (0), very high confidence (5), high confidence (4), moderate confidence (3), low confidence (2), very low or no confidence (1) Score=(Score to Q3+Score to Q4+Score to Q5+Score to Q6)x0.3
Mean Change from Baseline of "Lubrication" Score on the Female Sexual Function Index Questionnaire | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants answer questions:Q7. Over the past 4 weeks, how often did you become lubricated ("wet") during sexual activity or intercourse?Q9. Over the past 4 weeks, how often did you maintain your lubrication ("wetness") until completion of sexual activity or intercourse?Answers = Points: no sexual activity (0), almost always or always (5), most times (more than half the time) (4), sometimes (about half the time) (3), a few times (less than half the time) (2), almost never or never (1). Q8. Over the past 4 weeks, how difficult was it to become lubricated ("wet") during sexual activity or intercourse? Q10. Over the past 4 weeks, how difficult was it to maintain your lubrication ("wetness") until completion of sexual activity or intercourse? Answers = Points: no sexual activity (0), extremely difficult or impossible (1), very difficult (2), difficult (3), slightly difficult (4), not difficult (5). Score = (Score to Q7 + Score to Q8 + Score to Q9 + Score to Q10)x0.3
Mean Change from Baseline of "Orgasm" Score on the Female Sexual Function Index Questionnaire | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants answer questions:
  Q11. Over the past 4 weeks, when you had sexual stimulation or intercourse, how often did you reach orgasm (climax)? Answers = Points: no sexual activity (0), almost always or always (5), most times (4), sometimes (3), a few times (2), almost never or never (1).
  Q12. Over the past 4 weeks, when you had sexual stimulation or intercourse, how difficult was it for you to reach orgasm (climax)? Answers = Points: no sexual activity (0), extremely difficult or impossible (1), very difficult (2), difficult (3), slightly difficult (4), not difficult (5).
  Q13. Over the past 4 weeks, how satisfied were you with your ability to reach orgasm (climax) during sexual activity or intercourse? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Score = (Score to Q11 + Score to Q12 + Score to Q13)x0.4
Mean Change from Baseline of "Satisfaction" Score on the Female Sexual Function Index Questionnaire | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants answer questions:
  Q14. Over the past 4 weeks, how satisfied have you been with the amount of emotional closeness during sexual activity between you and your partner? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Q15. Over the past 4 weeks, how satisfied have you been with your sexual relationship with your partner? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Q16. Over the past 4 weeks, how satisfied have you been with your overall sexual life? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Score = (Score to Q14 + Score to Q15 + Score to Q16)x0.4
Mean Change from Baseline of "Pain" Score on the Female Sexual Function Index Questionnaire | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants answer questions:
  Q17. Over the past 4 weeks, how often did you experience discomfort or pain during vaginal penetration? Answers = Points: did not attempt intercourse (0), almost always or always (1), most times (2), sometimes (3), a few times (4), almost never or never (5).
  Q18. Over the past 4 weeks, how often did you experience discomfort or pain following vaginal penetration? Answers = Points: did not attempt intercourse (0), almost always or always (1), most times (2), sometimes (3), a few times (4), almost never or never (5).
  Q19. Over the past 4 weeks, how would you rate your level (degree) of discomfort or pain during or following vaginal penetration? Answers = Points: did not attempt intercourse (0)very high (1)high (2)moderate (3)low (4)very low or none at all (5).
  Score = (Score to Q17 + Score to Q18 + Score to Q19)x0.4
Mean Change from Baseline of Total Score on International Consultation on Incontinence Questionnaire - Short Form | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants answer questions:
  Q1 How often do you leak urine? Answers = Points: never (0), about once a week or less often (1), two or three times a week (2), about once a day (3), several times a day (4), all the time (5).
  Q2 How much urine do you usually leak? Answers = Points: none (0), a small amount (2), a moderate amount (4), a large amount (6) Q3 How much does leaking urine interfere with your everyday life? Answers = Visual Analogue Scale, where Not at all (0), A great deal (10).
  Total Score = Scores(Q1+Q2+Q3)
Mean Change from Baseline of "Physical Health Component Score" on The Short Form Health Survey | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants fill out a survey form (SF-36 Health Survey Standard Scoring). Calculations of final scores (PCS and MCS) will be carried out using Mean and SD from US adult population (PCS-US and MCS-US respectively).
Mean Change from Baseline of "Mental Health Component Score" on The Short Form Health Survey | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Participants fill out a survey form (SF-36 Health Survey Standard Scoring). Calculations of final scores (PCS and MCS) will be carried out using Mean and SD form US adult population (PCS-US and MCS-US respectively).
Mean Change from Baseline of pH of vagina | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Potential of hydrogen (pH) will be investigated by test-lines paper.
Mean Change from Baseline of Lactobacilli quantity | 1st visit (initial screening); 2nd visit (before the first treatment, no latter 2 months after 1st visit), 4th visit (before the last treatment, 8-12 weeks after 2nd visit); 5th visit (90 days after the last treatment - 4th visit)
  Smear will be sampled from the posterior wall of vagina and stained according to Gram. Evaluation of the Lactobacilli quantity will be performed for each participant with light microscope in field of view. Score depends on the number of bacteria: low - 1, average - 2, normal - 3.

CONTACTS AND LOCATIONS:
Overall Officials: Vladislav V Dubenskij, Ph.D., Principal Investigator — Tver State Medical Academy
Locations (1):
- Tver State Medical Academy, Tver', Tver Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
The following data can be shared with researchers upon an official request:
  The final version of the Study Protocol approved by the Local Ethics Committee; Copies of anonymized filled Individual Registration Cards (IRC); Informed Consent Form (ICF); Clinical Study Report (CSR) and/or published article (if not contradict the rules and conditions of a journal); Supplement files systematizing data.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD can be shared with researchers starting 3 months after CSR or article publication for five years.
Access Criteria: IPD can be shared with researchers only upon an official request from researcher's affiliation institution in the letter form on organization's letterhead paper signed by an authorized person. Official request must be directed by e-mail to the contact person (Ksenia Shatilova, shatilova@melsytech.com). The letter must contain the request purpose and statement of internal IPD use as confidential information only.
  IPD will be shared after approval by CEO of "MeLSyTech" Ltd according to the company internal rules. A requester will be notified of the decision by official letter. Depending on the decision, a requester will receive a link to the repository, or a justified rejection.